CLINICAL TRIAL: NCT04869475
Title: Arsenic Trioxide in Refractory Solid Tumors With Rescuable p53 Mutation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhang, Chief of department of oncology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANDA-Basket 1
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Refractory Solid Tumors
MeSH Terms: interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): arsenic trioxide 7mg/m2 ivgtt d1-14, q3w
  Interventions: Drug: Arsenic trioxide

INTERVENTIONS:
Drug: Arsenic trioxide — This is a single-arm study with all patients receiving arsenci trioxide.

SUMMARY:
This study is an open, prospective, single arm, multi center exploratory basket clinical study. 20 refractory solid tumors patients with rescuable p53 mutation will be enrolled, and the efficacy and safety of arsenic trioxide in those patients will be evaluated.

DETAILED DESCRIPTION:
p53 is the most frequently mutated protein in cancer. It is mutated in about half of all cancers and losses tumor-suppressive function. Yet there is no approved p53-targeted therapy, being one of the most unmet clinical needs. At least 45 approaches/agents were identified to kill cancer cells via p53 mutations by 2017, with at least 17 agents reported to function by restoring mutant p53 with wild-type p53 activity, yet these compounds are far from being able to achieve the desired outcome of converting all mutant p53 molecules to become fully'wild-type-like' .

In 2020, investigators reported the FDA-approved arsenic trioxide (ATO) as a mutant p53 rescue drug. Investigators firstly, based on the knowledge that the hundreds of p53 mutations inactivate p53 via heterogeneous mechanisms, proposed that there may be no single agent that is able to recue all of the'rainbow'p53 mutants. Investigators next proposed a rational mutant p53 rescue strategy, wherein the unfolded p53 mutants (termed as structural mutants) were precisely selected as rescue objects and, in addition, a thermostabilizing compounds were rationally used to promote the folding of structural mutants. Thirdly, investigators aimed at a cryptical completely-buried pocket inside p53 (in conventional targeted therapy, the targeted pockets are on the protein surface and thus exposed). By above, investigators identified ATO as a mutant p53 rescue compound, mechanistically mimicking the formation of disulfide bonds in C124-C135-C141 triad to promote the folding of structural mutants in the solved co-crystal structures (disulfide bond is one of the main forces to promote protein folding upon protein translation in classic biological chemistry textbook).

ATO differentiates itself from previously reported broad-spectrum mutant p53 rescue compounds in: (i) ATO is superior to the reported compounds by at least 100-time rescue efficiencies in promoting structural p53 mutants'thermostability, protein folding, specific DNA-binding ability, transcriptional activity, and other p53 activities in laboratories. (ii) the rescue is accompanied with a structural mechanism revealing how broad-spectrum p53 mutants (note: not all p53 mutants) can be rescued by a single small molecule. (iii) ATO is the compound that can only rescue a part of structural p53 mutations (it can not rescue all p53 mutations, it can not rescue all structural p53 mutations neither) and also a compound that has been experimentally applied and confirmed on dozens of p53 mutations.

ATO is the most effective APL leukemia treatment drug. When combined with ATRA, ATO cures APL leukemia (5-year survival from ~30% to over 90%). ATO was also reported to be efficacious in treating patients with non-APL hematological malignance and solid tumors, yet the response rate is low. Investigators thus proposed that it is p53 mutation conferring the treatment efficacy.

The hundreds of p53 mutations have wide-spectrum cancer distribution, and in addition, have highly diverse rescue efficiencies by ATO. Thus, cancer type selection and mutation selection are the two challenges in the current clinical trial (Note: These two challenges do not exist for the other targeted drugs such as the widely used EGFR inhibitors and the recent ground-breaking KRAS-G12C inhibitors since, according to the TCGA PanCancer Altas Studies, their applicable mutations predominately occur in one cancer type (both in lung adenocarcinoma), and clustered in one or few codons of their encoding genes). For these two challenges:

1. The current trial will focus on the cancer types predicted to highly dependent on p53 mutations, in other words, the p53 mutation should be a key driver in this cancer type and the cancer cells depend on the p53 mutation to survive and/or grow. Previous clinical trials have confirmed the importance of selecting appropriate cancer types for a targeted drug. For example, BRAFV600E inhibitors exhibit relatively high efficacy in treating BRAF-mutated melanoma, but not colorectal cancers.
2. The current trial will further precisely select p53 mutations that can be effectively and ideally, highly efficiently, rescued by ATO. Since ATO can only rescues a part of structural mutations, investigators thus initialized a large-scale project-PANDA (P53 AND Arsenic) cancer project since 2016, wherein investigators cloned the most frequent 800 p53 mutations individually (covering >95% p53 missense mutation cases in IARC) and quantified their rescue efficiencies by ATO for their transcriptional activities (the mutations were quantified individually), anti-proliferation ability in cancer cells, anti-tumor growth in xenograft mouse model, et al. In the PANDA cancer project, there is an apparent trend that ATO is most efficient in rescuing large-to-small amino acid mutations, mutations near the arsenic-binding pocket, temperature-sensitive mutations, as well as the mutations occurring on hydrophobic residues and in the LSH motif. Based on the rescue efficiencies by ATO, p53 mutations were stratified in several classes in the PANDA project (the open-access website for PANDA project is estimated to be completed in end of 2021). The patients harboring the class of p53 mutations that can be relatively efficiently and most efficiently rescued by ATO will be precisely recruited in the current trial.

The current exploratory trial was termed as PANDA-bascket1.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patients aged≥18 years.
2. Patients with refractory solid tumors were confirmed by histopathology and structural p53 mutations were confirmed by sanger sequence.
3. ECOG performance status 0 or 2, expected lifetime≥3 months.
4. Adequate organ function: Absolute neutrophil count (ANC) ≥1.5x109/L, White blood count ≥3.5x109/L, Platelets ≥75x109/L, Hemoglobin (Hb) ≥70g/L, ALT/AST ≤2.5x ULN (for patient with liver metastasis ALT/AST ≤5x ULN), Serum bilirubin ≤1.5x ULN, Serum creatinine ≤1.5x ULN.
5. HBV infected patients (inactive/asymptomatic carrier, chronic or active) with HBV DNA<500IU/ml (or 2500 copies/ml).
6. Pregnancy test of female patients with fertile activity should be negative within 7 days before enrollment. Patients should keep contraception during treatment.
7. Willingness and ability to comply with the protocol for the duration of the study including scheduled visits, examinations, investigations and treatment plans with informed consent form.

Exclusion Criteria:

1. Pregnancy or children bearing potential.
2. brain or meningeal metastasis.
3. With second primary malignant diseases.
4. With uncontrolled auto-immune diseases, interstitial pneumonia, ulcerative colitis, or patients who should receive long-term glucocorticoid treatment (>10mg/d prednisone).
5. With uncontrollable complications
6. Inadequate organ function
7. Conditions which impact on pill taking (dysphagia, chronic diarrhea, bowel obstruction).
8. known hypersensitivity reaction to any of the study drugs or components.
9. Other unsuitable conditions determined by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) | 12 months

SECONDARY OUTCOMES:
Overall response rate (ORR) | 12 months
Progression free survival (PFS) | 12 months
Duration of response (DOR) | 12 months
Safety: adverse events as assessed by CTCAE v5.0 | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Min Lu, Ph. D, Principal Investigator — Ruijin Hospital; Jun Zhang, MD & PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Department of Oncology, Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canon J, Rex K, Saiki AY, Mohr C, Cooke K, Bagal D, Gaida K, Holt T, Knutson CG, Koppada N, Lanman BA, Werner J, Rapaport AS, San Miguel T, Ortiz R, Osgood T, Sun JR, Zhu X, McCarter JD, Volak LP, Houk BE, Fakih MG, O'Neil BH, Price TJ, Falchook GS, Desai J, Kuo J, Govindan R, Hong DS, Ouyang W, Henary H, Arvedson T, Cee VJ, Lipford JR. The clinical KRAS(G12C) inhibitor AMG 510 drives anti-tumour immunity. Nature. 2019 Nov;575(7781):217-223. doi: 10.1038/s41586-019-1694-1. Epub 2019 Oct 30. PMID 31666701
- [Background] Chen S, Wu JL, Liang Y, Tang YG, Song HX, Wu LL, Xing YF, Yan N, Li YT, Wang ZY, Xiao SJ, Lu X, Chen SJ, Lu M. Arsenic Trioxide Rescues Structural p53 Mutations through a Cryptic Allosteric Site. Cancer Cell. 2021 Feb 8;39(2):225-239.e8. doi: 10.1016/j.ccell.2020.11.013. Epub 2020 Dec 24. PMID 33357454
- [Background] Kopetz S, Desai J, Chan E, Hecht JR, O'Dwyer PJ, Maru D, Morris V, Janku F, Dasari A, Chung W, Issa JP, Gibbs P, James B, Powis G, Nolop KB, Bhattacharya S, Saltz L. Phase II Pilot Study of Vemurafenib in Patients With Metastatic BRAF-Mutated Colorectal Cancer. J Clin Oncol. 2015 Dec 1;33(34):4032-8. doi: 10.1200/JCO.2015.63.2497. Epub 2015 Oct 12. PMID 26460303
- [Background] Sabapathy K, Lane DP. Therapeutic targeting of p53: all mutants are equal, but some mutants are more equal than others. Nat Rev Clin Oncol. 2018 Jan;15(1):13-30. doi: 10.1038/nrclinonc.2017.151. Epub 2017 Sep 26. PMID 28948977
- [Background] Wang H, Liu Y, Wang X, Liu D, Sun Z, Wang C, Jin G, Zhang B, Yu S. Randomized clinical control study of locoregional therapy combined with arsenic trioxide for the treatment of hepatocellular carcinoma. Cancer. 2015 Sep 1;121(17):2917-25. doi: 10.1002/cncr.29456. Epub 2015 May 29. PMID 26033499
- [Background] Zhang TD, Chen GQ, Wang ZG, Wang ZY, Chen SJ, Chen Z. Arsenic trioxide, a therapeutic agent for APL. Oncogene. 2001 Oct 29;20(49):7146-53. doi: 10.1038/sj.onc.1204762. PMID 11704843
- [Derived] Tang Y, Song H, Wang Z, Xiao S, Xiang X, Zhan H, Wu L, Wu J, Xing Y, Tan Y, Liang Y, Yan N, Li Y, Li J, Wu J, Zheng D, Jia Y, Chen Z, Li Y, Zhang Q, Zhang J, Zeng H, Tao W, Liu F, Wu Y, Lu M. Repurposing antiparasitic antimonials to noncovalently rescue temperature-sensitive p53 mutations. Cell Rep. 2022 Apr 12;39(2):110622. doi: 10.1016/j.celrep.2022.110622. PMID 35417717